CLINICAL TRIAL: NCT05366608
Title: 14.0- 3.0- 3.0- η Protein is Associated With Disease Activity and Osteoporosis in Patients With Rheumatoid Arthritis
Brief Title: 14.0- 3.0- 3.0- η Protein With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.21.11.1528 - 2021/11/21
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Disease Activity
Keywords: Rheumatoid arthritis; osteoporosis; 14.0- 3.0- 3.0- η
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients: 188 patients with RA he RA activity parameters were evaluated in RA patients. BMD was measured. Serum level of 14.0- 3.0- 3.0- η protein and IL_.6 were estimated for all participants by ELISA.
  Interventions: Diagnostic Test: Serum level of 14.0- 3.0- 3.0- η protein and IL_.6
- Control: 192 matched controls were enrolled. T
  Interventions: Diagnostic Test: Serum level of 14.0- 3.0- 3.0- η protein and IL_.6

INTERVENTIONS:
Diagnostic Test: Serum level of 14.0- 3.0- 3.0- η protein and IL_.6 — Serum level of 14.0- 3.0- 3.0- η protein and IL_.6 were estimated for all participants by ELISA.
  Other Names: ELISA

SUMMARY:
Aim of work: to explore the potential association between serum 14.0-3.0-3.0- η protein level with disease activity and bone mineral density (BMD) in Egyptian patients with rheumatoid arthritis (RA).

188 patients with RA and 192 matched controls were enrolled. The RA activity parameters were evaluated in RA patients. BMD was measured. Serum level of 14.0- 3.0- 3.0- η protein and IL_.6 were estimated for all participants by ELISA.

DETAILED DESCRIPTION:
A total of 200 RA patients were invited to be enrolled in this study. Patients were diagnosed as having RA by the 2010 European-league-against-Rheumatism- (EULAR) and American-College-of-rheumatology (ACR) classification criteria for RA. Patients were collected from the outpatient clinic of the Rheumatology and Rehabilitation Department, Mansoura University Hospital.

All participants underwent detailed medical history taking as well as clinical examination. The medical records of all patients were carefully reviewed. Data collection included age, gender, past medical history, current and past drug intake. In RA patients, the disease duration, duration of the morning stiffness, tender joint count (TJC) and swollen joint count (SJC) were reported. The activity of RA was measured by disease activity score 28 (DAS.28) based on the erythrocyte sedimentation rate (ESR) level (DAS28-ESR) [19]. The intensity of perceived pain was assessed by the visual analog scale (VAS) 100-mm scale.

Bone mineral density (BMD) was measured using dual energy X-ray absorptiometry (DEXA) at proximal femur for all participants who were categorized into normal, osteopenic, or osteoporotic according to the definition of the World Health Organization (WHO) of the recorded T score A commercially available human IL_.6 ELISA kit (GenProbe, Diaclone, France) was used to measure IL_.6 serum level following the instructions of the manufacturer.

Serum level of 14.0- 3.0- 3.0- η protein was determined by ELISA for all participants,

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as having RA by the 2010 European-league-against-Rheumatism- (EULAR) and American-College-of-rheumatology (ACR) classification criteria for RA Patients were collected from the outpatient clinic of the Rheumatology and Rehabilitation Department, Mansoura University Hospital

Exclusion Criteria:

* postmenopausal females, patients with other rheumatic autoimmune diseases, severe infection, diabetes mellitus, hypertension, liver or kidney disease, malignancies, endocrinal diseases, pregnant or lactating females. Patients with current intake of glucocorticoids, anticonvulsants, estrogen or anti-coagulant, alcohol users, or other factors that lead to secondary osteoporosis were also excluded from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: RA patients were invited to be enrolled in this study. Patients were diagnosed as having RA by the 2010 European-league-against-Rheumatism- (EULAR) and American-College-of-rheumatology (ACR) classification criteria for RA
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
primary | 2 years
  potential association between serum 14.0-3.0-3.0- η protein level with disease activity

SECONDARY OUTCOMES:
secondry | 2 years
  association between serum 14.0-3.0-3.0- η protein level with bone mineral density (BMD)

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin A Abdelsalam, MD, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided